CLINICAL TRIAL: NCT04019860
Title: Isolated and Combined Effects of High Intensity Interval Training and Time Restricted Eating on Glycaemic Control in Reproductive-aged Women With Overweight or Obesity
Brief Title: Time-restricted Eating and High Intensity Interval Training Among Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Australian Catholic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2019/851; 285171 (Other: Comittee for Medical and Health Research Ethics Mid Norway)
Record Dates: First submitted 2019-07-09; First posted 2019-07-15 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: Obesity; Endocrine
Keywords: Exercise; Diet; Overweight; Glycaemic control; Fitness; Body composition
MeSH Terms: conditions — Obesity; Motor Activity; Overweight | interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: Four-armed randomised controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- High Intensity Interval Training (Experimental): High intensity interval training for seven weeks. Three weekly, supervised training sessions.
  Interventions: Behavioral: High Intensity Interval Training
- Time-Restricted Eating (Experimental): Time-restricted eating for seven weeks. Maximal daily eating window of 10 hours.
  Interventions: Behavioral: Time-Restricted Eating
- High Intensity Interval Training & Time-Restricted Eating (Experimental)
  Interventions: Behavioral: High Intensity Interval Training; Behavioral: Time-Restricted Eating
- Control (No Intervention): Will be given information about the recommended level of physical activity for health benefits and a healthy diet.

INTERVENTIONS:
Behavioral: High Intensity Interval Training — Three weekly, supervised exercise sessions with high intensity. Each session will last for 30-45 minutes. Intervention period will be seven weeks.
  Arms: High Intensity Interval Training; High Intensity Interval Training & Time-Restricted Eating
Behavioral: Time-Restricted Eating — Restricted daily window of caloric intake to maximum 10 hours. Intervention period will be seven weeks.
  Arms: High Intensity Interval Training & Time-Restricted Eating; Time-Restricted Eating

SUMMARY:
This project will determine the independent and combined effects of high intensity interval training and time-restricted eating on blood sugar regulation among women in reproductive-age who have overweight or obesity. The intervention period will be seven weeks. Before and after the intervention, blood sugar regulation, body composition and physical fitness will be measured and compared between groups who are doing either high intensity interval training, time-restricted eating, both high intensity interval training and time-restricted eating, or who are in a control group. Physical activity, sleep quality, continuous glucose monitoring, adherence to the interventions and hunger/satiety will also be measured.

DETAILED DESCRIPTION:
In a follow-up study, we will invite randomized participants to come in for new assessments of physical fitness, body composition and fasting blood samples, and they will be asked to complete questionnaires about adherence to the interventions two years after intervention-end. The first participants will come in to the laboratory for the two-year follow up in November 2021.

ELIGIBILITY:
Inclusion Criteria:

* body mass index ≥ 27 kg/cm2,
* able to walk on a treadmill or ride a bike for at least 60 min.

Exclusion Criteria:

* Pregnancy, lactation within 24 weeks of study commencement
* known cardiovascular disease
* type 1 or 2 diabetes
* currently taking hypertension or glucose- or lipid-lowering medication
* habitual eating window < 12 hours
* performing high intensity training more than once a week
* body mass variations > 4 kg three months prior to study commencement
* shift work that includes night shifts.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 131 (Actual)
Dates: Start 2019-08-12 (Actual); Primary Completion 2021-03-16 (Actual); Study Completion 2021-03-16 (Actual)

PRIMARY OUTCOMES:
Glycaemic control | From baseline to after 7 weeks intervention
  Total area under the plasma glucose curve over two hours after a 75 g oral glucose tolerance test

SECONDARY OUTCOMES:
Insulin sensitivity | From baseline to after 7 weeks intervention
  Insulin sensitivity estimated by homeostatic model assessment for insulin resistance (fasting serum insulin concentration (μU/mL) x fasting plasma glucose levels (mmol/L)/22.5)
Insulin levels after ingestion of glucose | From baseline to after 7 weeks intervention
  Total area under the serum insulin two hours after a 75 g oral glucose tolerance test
Cardiorespiratory fitness | From baseline to after 7 weeks intervention
  Peak oxygen uptake at a maximum effort exercise test, measured in mL/min/kg and L/min
Body mass | From baseline to after 7 weeks intervention
  In kg
Body fat mass | From baseline to after 7 weeks intervention
  In kg
Body fat percentage | From baseline to after 7 weeks intervention
  In percent of total body mass
Fat-free body mass | From baseline to after 7 weeks intervention
  In kg
Fat-free body mass percentage | From baseline to after 7 weeks intervention
  In percent of total body mass
Systolic blood pressure | From baseline to after 7 weeks intervention
  Average of three measurements, in mmHg
Diastolic blood pressure | From baseline to after 7 weeks intervention
  Average of three measurements, in mmHg
Resting heart rate | From baseline to after 7 weeks intervention
  Average of three measurements, in beats/min
Cholesterol in blood | From baseline to after 7 weeks intervention
  Total fasting cholesterol in blood
High density lipoprotein cholesterol in blood | From baseline to after 7 weeks intervention
  Fasting high density lipoprotein cholesterol i blood
Low density lipoprotein cholesterol in blood | From baseline to after 7 weeks intervention
  Fasting low density lipoprotein cholesterol i blood
Triglycerides in blood | From baseline to after 7 weeks intervention
  Fasting low density lipoprotein cholesterol i blood
Average glucose levels | From baseline to after 7 weeks intervention
  Glycated haemoglobin (HbA1c)
Insulinemia | From baseline to after 7 weeks intervention
  Fasting insulin in blood
24 hour glycaemic control | From baseline to the last 14 days of the intervention period
  Average interstitial glucose levels during 24 h, area under the curve
Postprandial glycaemic control | From baseline to the last 14 days of the intervention period
  Average interstitial glucose levels 3 hours after the first meal of the day, area under the curve
Nocturnal glycaemic control | From baseline to the last 14 days of the intervention period
  Average interstitial glucose levels from 23:00 h to 06:00 h
Self-reported physical activity | From baseline to after 7 weeks intervention
  International Physical Activity Questionnaire
Measured physical activity | From baseline to the last 14 days of the intervention period
  Measure by Sensewear activity monitor
Sleep | From baseline to after 7 weeks intervention
  Self-reported: Pittsburgh Sleep Quality Index
Chronotype | From baseline to after 7 weeks intervention
  Self-reported: Hornestberg Morningness Eveningness Questionnaire

OTHER OUTCOMES:
Adherence to high intensity interval training | Seven weeks
  Number of completed exercise sessions out of those prescribed, in percentage
Compliance to high intensity interval training | Seven weeks
  Exercise intensity, heart rate in percentage of individual heart rate maximum
Compliance to time-restricted eating | Seven weeks
  Average daily eating window, in hours
Adherence to time-restricted eating | Seven weeks
  Average number of days where per week that daily eating window is 10 hours or less.
Diet intake at baseline | 14 days at baseline (one week of habitual diet and one week after the intervention starts)
  Online food diary
Diet intake | The last 14 days of the intervention
  Online food diary

CONTACTS AND LOCATIONS:
Overall Officials: Øystein T Risa, PhD, Study Director — Norwegian University of Science and Technology; Trine T Moholdt, PhD, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- Department of circulation and medical imaging , NTNU, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Haganes KL, Devlin BL, Orr RK, Moholdt T. Impact of Time-Restricted Eating and High-Intensity Exercise on Nutrient Intake in Women with Overweight/Obesity: Secondary Analysis of a Randomized Controlled Trial. Nutrients. 2025 Jan 8;17(2):218. doi: 10.3390/nu17020218. PMID 39861348
- [Derived] Haganes KL, Silva CP, Eyjolfsdottir SK, Steen S, Grindberg M, Lydersen S, Hawley JA, Moholdt T. Time-restricted eating and exercise training improve HbA1c and body composition in women with overweight/obesity: A randomized controlled trial. Cell Metab. 2022 Oct 4;34(10):1457-1471.e4. doi: 10.1016/j.cmet.2022.09.003. PMID 36198292
- [Derived] Moholdt T, Silva CP, Lydersen S, Hawley JA. Isolated and combined effects of high-intensity interval training and time-restricted eating on glycaemic control in reproductive-aged women with overweight or obesity: study protocol for a four-armed randomised controlled trial. BMJ Open. 2021 Feb 5;11(2):e040020. doi: 10.1136/bmjopen-2020-040020. PMID 33550228